CLINICAL TRIAL: NCT03118050
Title: Identifying Therapeutic Targets of Accelerated Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 15-0229/17-0064; R01AG049611 (NIH)
Record Dates: First submitted 2016-12-08; First posted 2017-04-18 (Actual); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Sarcopenia; Diabetes Mellitus; Aging
Keywords: exercise; bed rest; muscle; nutrition; amino acids
MeSH Terms: conditions — Sarcopenia; Diabetes Mellitus; Motor Activity | interventions — Resistance Training; Bed Rest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- RT in T2DM (Experimental): Type 2 diabetes subjects will undergo 3 months of resistance exercise training. Muscle size, strength and response to a low dose amino acids will be measured before and after training. Results of this arm will be compared to those previously obtained in healthy older subjects who participated in NCT02999802 (same training protocol) after 1:1 matching for age and sex.
  Interventions: Behavioral: Resistance exercise training
- BR in healthy subjects, LAA (Experimental): Healthy subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Interventions: Behavioral: Bed rest
- BR in healthy subjects, HAA (Experimental): Healthy subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a high dose amino acids (HAA) will be measured before and after bed rest.
  Interventions: Behavioral: Bed rest
- BR in T2DM, LAA (Experimental): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Interventions: Behavioral: Bed rest
- BR in T2DM, HAA (Experimental): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a high dose amino acids (HAA) will be measured before and after bed rest.
  Interventions: Behavioral: Bed rest
- BR in healthy subjects, PT (Experimental): Healthy subjects will undergo short term bed rest with intensive physical therapy (PT). Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Interventions: Behavioral: Bed rest; Behavioral: Intensive physical therapy
- BR in T2DM, PT (Experimental): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with intensive physical therapy (PT). Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Interventions: Behavioral: Bed rest; Behavioral: Intensive physical therapy

INTERVENTIONS:
Behavioral: Resistance exercise training — Supervised resistance exercise training, 3 times a week for 3 months
  Other Names: RT
  Arms: RT in T2DM
Behavioral: Bed rest — Bed rest for 5 days, followed by standard rehabilitation for 2 days
  Other Names: BR
  Arms: BR in T2DM, HAA; BR in T2DM, LAA; BR in T2DM, PT; BR in healthy subjects, HAA; BR in healthy subjects, LAA; BR in healthy subjects, PT
Behavioral: Intensive physical therapy — Intensive weight bearing PT, daily, during bed rest
  Other Names: PT
  Arms: BR in T2DM, PT; BR in healthy subjects, PT

SUMMARY:
The proposed research is designed to identify the mechanisms that can accelerate loss of muscle size, strength and physical function in type 2 diabetes and with hospitalization in older persons. About ⅓ of older Americans have type 2 diabetes, and about ⅓ of the hospitalizations in the USA involve persons older than 65 year of age. The proposed research is relevant to the part of NIH's mission that pertains to development of the fundamental knowledge that will improve health and reduce the burdens of disability, because this work will provide the fundamental evidence to identify new targets for the development of innovative treatments to slow down muscle loss and disability in our aging society.

DETAILED DESCRIPTION:
Sarcopenia is a major contributor to frailty and increases the risk of falls, physical dependence, disability and mortality in older adults. It advances slowly with healthy aging. However, diseases or other insults and injuries can accelerate sarcopenia and lead to catastrophic declines in mobility and independence. For example, chronic diseases such as Type 2 Diabetes Mellitus (T2DM) are associated with accelerated loss of muscle mass and function in seniors; hospitalization with bed rest inactivity acutely accelerates sarcopenia. What it is not known is how concurrent diseases, inactivity or other insults and injuries accelerate sarcopenia in older adults. This knowledge gap hinders the development of innovative, targeted treatments for this disabling condition. The objective of this research is to examine the basic mechanisms that underlie accelerated sarcopenia in older adults and identify potential targets for interventions. The central hypothesis is that a global and fundamental mechanism of acute or chronic acceleration of sarcopenia is a reduction in skeletal muscle amino acid transport, which decreases muscle protein anabolism, and can be reversed by activation of the mammalian/mechanistic Target of Rapamycin Complex 1 (mTORC1) signaling with a non-amino acid stimulus, such as exercise. Amino acid transport is an active process that controls intracellular amino acid availability and the activation of protein synthesis in skeletal muscle. It is regulated by amino acid concentrations and non-amino acid stimuli that activate mTORC1 signaling, such as resistance exercise and insulin.The central hypothesis will be tested with the following specific aims: 1) Determine the effect of T2DM on the sensitivity of skeletal muscle amino acid transport to dietary amino acids. 2) Determine the effect of short-term bed rest inactivity on the sensitivity of skeletal muscle amino acid transport to dietary amino acids. 3) Determine the effect of resistance exercise on the sensitivity of amino acid transport to dietary amino acids in acute and chronic accelerated sarcopenia induced by inactivity or T2DM. Amino acid transport and protein metabolism in muscle will be measured using integrative molecular, imaging and stable isotope methodologies, identifying specific upstream regulators involved in the anabolic resistance of accelerated sarcopenia that can be targeted with novel treatments to reduce sarcopenia and improve independence in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index: <40 kg/sq meter
* Score ≥26 on the 30-item Mini Mental State Examination
* Stable body weight for at least 3 months
* Non-diabetic or with Type 2 Diabetes Mellitus

Exclusion Criteria:

* Pre-diabetes per American Diabetes Association criteria
* Insulin therapy, significant diabetic complications, or A1c>8%
* Impairment in Activities of Daily Living
* >2 falls/year
* weight loss >5% in the past 6 months
* Exercise training (≥2 sessions/week) or ≥10,000 steps/day
* Significant cardiovascular, liver, renal, blood, or respiratory disease
* Active cancer or infection
* Recent (within 3 months) treatment with anabolic steroids, systemic corticosteroids or estrogen.
* Alcohol or drug abuse

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-05-28 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Volpi, MD, PhD, Principal Investigator — UTMB
Locations (1):
- Sealy Center on Aging, University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Small physiological study. Few subjects. Risk of loss of confidentiality

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were randomized to one of six bed rest (BR) study arms under IRB protocol 17-0064. Separately, eligible participants were randomized to one of six resistance training (RT) study arms under IRB protocol 15-0229. The RT data were analyzed in comparison with de-identified data obtained from NTC02999802.
Groups:
- Resistance Training in Type 2 Diabetes (T2DM): Type 2 diabetes subjects will undergo 3 months of resistance exercise training. Muscle size, strength and response to a low dose amino acids will be measured before and after training. Results of this arm will be compared to those previously obtained in healthy older subjects who participated in NCT02999802 (same training protocol) after 1:1 matching for age and sex.
  Resistance exercise training: Supervised resistance exercise training, 3 times a week for 3 months
- Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA): Healthy subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days. UTMB IRB 17-0064
- Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA): Healthy subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a high dose amino acids (HAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days. UTMB IRB 17-0064
- Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days
- Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a high dose amino acids (HAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days
- Bed Rest in Healthy Subjects, Physical Therapy (PT): Healthy subjects will undergo short term bed rest with intensive physical therapy (PT). Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days
  Intensive physical therapy: Intensive weight bearing PT, daily, during bed rest. UTMB IRB 17-0064
- BR in T2DM, PT: Type 2 diabetes (T2DM) subjects will undergo short term bed rest with intensive physical therapy (PT). Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days
  Intensive physical therapy: Intensive weight bearing PT, daily, during bed rest. UTMB IRB 17-0064
Period: Overall Study
Arm/Group | Resistance Training in Type 2 Diabetes (T2DM) | Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) | Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) | Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) | Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) | Bed Rest in Healthy Subjects, Physical Therapy (PT) | BR in T2DM, PT
Started | 29 | 12 | 11 | 11 | 9 | 12 | 11
Completed | 15 | 7 | 5 | 6 | 5 | 6 | 6
Not Completed | 14 | 5 | 6 | 5 | 4 | 6 | 5
Not completed — Did not meet inclusion criteria after signing consent form | 14 | 5 | 6 | 5 | 4 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA): Healthy subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a high dose amino acids (HAA) will be measured. before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days. UTMB IRB 17-0064
- Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days. UTMB IRB 17-0064
- Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with standard of care physical therapy. Muscle size, strength and response to a high dose amino acids (HAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days. UTMB IRB 17-0064
- Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with intensive physical therapy (PT). Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days
  Intensive physical therapy: Intensive weight bearing PT, daily, during bed rest. UTMB IRB 17-0064
- Total: Total of all reporting groups
Arm/Group | Resistance Training in Type 2 Diabetes (T2DM) | Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) | Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) | Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) | Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) | Bed Rest in Healthy Subjects, Physical Therapy (PT) | Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT) | Total
Number analyzed (Participants) | 15 | 7 | 5 | 6 | 5 | 6 | 6 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (4) | 67 (7) | 73 (6) | 70 (5) | 71 (8) | 64 (1) | 68 (6) | 69 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 2 | 4 | 3 | 4 | 4 | 27
  Male | 10 | 2 | 3 | 2 | 2 | 2 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 6
  Not Hispanic or Latino | 13 | 6 | 4 | 5 | 4 | 6 | 6 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 5
  White | 14 | 6 | 4 | 6 | 4 | 6 | 5 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 5 | 6 | 5 | 6 | 6 | 50

OUTCOME MEASURES:

1. Primary Outcome: Leg Lean Mass
Description: Measurement of change in leg lean mass by DEXA
Time Frame: Change from baseline to up to 3 months
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT): Type 2 diabetes (T2DM) subjects will undergo short term bed rest with intensive physical therapy (PT). Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days
  Intensive physical therapy: Intensive weight bearing PT, daily, during bed rest. UTMB 17-0064
Arm/Group | Resistance Training in Type 2 Diabetes (T2DM) | Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) | Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) | Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) | Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) | Bed Rest in Healthy Subjects, Physical Therapy (PT) | Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT)
Number analyzed (Participants) | 15 | 7 | 5 | 6 | 5 | 6 | 6
kg | 0.35 (0.74) | -0.55 (0.42) | -0.80 (0.44) | -0.44 (0.32) | -0.66 (0.31) | -0.59 (0.73) | -0.40 (0.34)
Statistical Analysis 1: Comparison: Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) vs Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) vs Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) vs Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) vs Bed Rest in Healthy Subjects, Physical Therapy (PT) vs Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT); Test type: Other; p < 0.01, ANOVA — Main effect of bed rest

2. Secondary Outcome: Knee Extension Strength
Description: Measurement of change in maximum strength by standard method
Time Frame: Change from baseline to up to 3 months
Measure: Mean (Standard Deviation); unit: Nm
Arm/Group | Resistance Training in Type 2 Diabetes (T2DM) | Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) | Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) | Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) | Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) | Bed Rest in Healthy Subjects, Physical Therapy (PT) | Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT)
Number analyzed (Participants) | 15 | 7 | 5 | 6 | 5 | 6 | 6
Nm | 3 (11) | -12 (20) | -24 (16) | -23 (13) | -30 (14) | -14 (9) | -8 (22)
Statistical Analysis 1: Comparison: Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) vs Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) vs Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) vs Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) vs Bed Rest in Healthy Subjects, Physical Therapy (PT) vs Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT); Test type: Other; p < 0.01, ANOVA — Main effect of bed rest

3. Other Pre Specified Outcome: Amino Acid Transporter Expression
Description: Measurement of change in amino acid transporter expression
Time Frame: Change from baseline to up to 3 months
Reporting Status: Not Posted, anticipated posting 2026-10

4. Other Pre Specified Outcome: Muscle Protein Synthesis
Description: Measurement of change in muscle protein synthesis by standard stable isotope methodology
Time Frame: Change from baseline to up to 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from baseline through 1 week following completion of the intervention period.
Groups:
- Bed Rest in Healthy Subjects, Physical Therapy (PT)Subjects, PT: Healthy subjects will undergo short term bed rest with intensive physical therapy (PT). Muscle size, strength and response to a low dose amino acids (LAA) will be measured before and after bed rest.
  Bed rest: Bed rest for 5 days, followed by standard rehabilitation for 2 days
  Intensive physical therapy: Intensive weight bearing PT, daily, during bed rest. UTMB IRB 17-0064
Arm/Group | Resistance Training in Type 2 Diabetes (T2DM) | Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) | Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) | Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) | Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) | Bed Rest in Healthy Subjects, Physical Therapy (PT)Subjects, PT | Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7 | 1/5 | 0/6 | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7 | 0/5 | 0/6 | 0/5 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/15 | 0/7 | 0/5 | 0/6 | 0/5 | 0/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resistance Training in Type 2 Diabetes (T2DM) (N=15) | Bed Rest in Healthy Subjects, Low-dose Amino Acids (LAA) (N=7) | Bed Rest in Healthy Subjects, High-dose Amino Acids (HAA) (N=5) | Bed Rest in Type 2 Diabetes (T2DM), Low-dose Amino Acids (LAA) (N=6) | Bed Rest in Type 2 Diabetes (T2DM), High-dose Amino Acids (HAA) (N=5) | Bed Rest in Healthy Subjects, Physical Therapy (PT)Subjects, PT (N=6) | Bed Rest in Type 2 Diabetes (T2DM), Physical Therapy (PT) (N=6)
Home medication error (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) — The participant accidentally took a double dose of prescribed blood pressure medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol: 15-0229 Study Protocol (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/50/NCT03118050/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: 17-0064 Study Protocol (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT03118050/Prot_SAP_001.pdf